CLINICAL TRIAL: NCT04094818
Title: TriVerity in the Diagnosis and Prognosis of Emergency Department Patients With Suspected Infections and Suspected Sepsis
Acronym: SEPSIS-SHIELD
Status: Completed | Type: Observational
Sponsor: Inflammatix (Industry)
Responsible Party: Sponsor
Other Study IDs: INF-04
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections; Intra-Abdominal Infections; Skin and Soft Tissue Infection; Suspected Meningitis/Encephalitis or Any Other Infection; Sepsis
Keywords: Infection; mRNA; Procalcitonin; C-Reactive Protein; Lactate
MeSH Terms: conditions — Respiratory Tract Infections; Urinary Tract Infections; Intraabdominal Infections; Soft Tissue Infections; Encephalitis; Sepsis; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PAXgene RNA tubes containing whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TriVerity — Blood collection for mRNA analysis, Procalcitonin and CRP determination, molecular analysis of nasopharyngeal swab collection and sputum/ BAL sample collection
  Other Names: InSep; HostDx Sepsis

SUMMARY:
This study will analyze gene expression and other laboratory data from biological samples collected from participants with suspected respiratory, urinary, intra-abdominal, and/or skin & soft tissue infections; or suspected sepsis of any cause.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 year
2. Suspected acute infection (respiratory, urinary, abdominal, skin & soft-tissue), and at least one of the symptoms OR, Suspected sepsis of any cause as defined by a blood culture order by the treating physician, and at least two of the symptoms:

   * Heart rate: >90 beats/ minute
   * Temperature: >38 C or <36C
   * Respiratory Rate: >20 breaths / minutes or PaO2 of <60 mmHg or SpO2 <90%
   * Systolic blood pressure: <100 mmHg
   * Altered mental status: Per clinical exam
3. Able to provide informed consent, or consent by legally authorized representative.

Exclusion Criteria:

Participants will be ineligible for this study if they meet any of the following criteria:

1. Patient-reported treatment with systemic antibiotics, systemic antiviral agents or systemic antifungal agents within the past 7 days prior to the emergency department study visit. Participants will not be excluded for use of:

   1. Antiviral treatment for HIV infection and hepatitis B and hepatitis C
   2. Topical antibiotics, topical antiviral or topical antifungal agents
   3. Anti-herpes prophylaxis aiding suppression of a recuring herpes infection
   4. Peri-operative (prophylactic) antibiotics
   5. A single dose of antimicrobials during the present ED visit (<10h before blood draw); note single dose can be considered mono or combination therapy, wherein combination is administered as part of local Standard of Care and only one dose of each medication is administered within the allowable 10-hour window
2. Patients receiving palliative or hospice care, or those receiving limited interventional care.
3. Prisoners, mentally disabled, or unable to give consent. Should the patient not be able to provide informed consent the legally authorized representative can provide the consent on behalf of the patient.
4. Patients receiving experimental therapy or already enrolled in an interventional clinical trial in which a subject receives some type of intervention, which can include but is not limited to investigational drugs, medical devices, or vaccines.

   a. Subjects that are enrolled in non-interventional or observational clinical trials will be allowed to participate in this clinical trial.
5. Patients previously enrolled in the present clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency departments of enrolling sites with:
  1. Suspected infection and one or more abnormal vital signs, OR
  2. Patients with suspected sepsis of any cause as defined by a blood culture order by the treating physician and two or more abnormal vital signs
Sampling Method: Non-Probability Sample
Enrollment: 1441 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the diagnostic performance of HostDx Sepsis | 28 Days After Enrollment
  Concordance of HostDx Sepsis bacterial readout with clinical adjudication
Evaluation of the diagnostic performance of HostDx Sepsis | 28 Days After Enrollment
  Concordance of HostDx Sepsis viral readout with clinical adjudication
Evaluation of the prognostic performance of HostDx Sepsis | 7 Days After Enrollment
  Concordance of HostDx Sepsis severity readout with receipt of ICU-level care (including requirement for ICU transfer, mechanical ventilation, vasopressors, or renal replacement therapy (RRT))

SECONDARY OUTCOMES:
Evaluation of the prognostic performance of HostDx Sepsis | 28 Days after enrollment
  Concordance of HostDx Sepsis severity readout with receipt of ICU-level care (including requirement for ICU transfer, mechanical ventilation, vasopressors, or renal replacement therapy (RRT)) within 7 days OR 28-Day Hospital Mortality
Evaluation of the prognostic performance of HostDx Sepsis for 28-Day Hospital Mortality | 28 Days after enrollment
  Concordance of HostDx Sepsis severity readout with 28-Day Hospital Mortality

CONTACTS AND LOCATIONS:
Locations (26):
- United States (25):
  - University of South Alabama, Mobile, Alabama
  - University of Southern California, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - University of Florida (UF) - Jacksonville, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Hackensack Meridian Health, Montclair, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma University Health, Oklahoma City, Oklahoma
  - Geisinger Health, Danville, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center - El Paso, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- ATTIKON University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaieski DF, Mikkelsen ME, Band RA, Pines JM, Massone R, Furia FF, Shofer FS, Goyal M. Impact of time to antibiotics on survival in patients with severe sepsis or septic shock in whom early goal-directed therapy was initiated in the emergency department. Crit Care Med. 2010 Apr;38(4):1045-53. doi: 10.1097/CCM.0b013e3181cc4824. PMID 20048677
- [Background] Ferrer R, Martin-Loeches I, Phillips G, Osborn TM, Townsend S, Dellinger RP, Artigas A, Schorr C, Levy MM. Empiric antibiotic treatment reduces mortality in severe sepsis and septic shock from the first hour: results from a guideline-based performance improvement program. Crit Care Med. 2014 Aug;42(8):1749-55. doi: 10.1097/CCM.0000000000000330. PMID 24717459
- [Background] Mi MY, Klompas M, Evans L. Early Administration of Antibiotics for Suspected Sepsis. N Engl J Med. 2019 Feb 7;380(6):593-596. doi: 10.1056/NEJMclde1809210. No abstract available. PMID 30726686
- [Background] Singer M. Biomarkers in sepsis. Curr Opin Pulm Med. 2013 May;19(3):305-9. doi: 10.1097/MCP.0b013e32835f1b49. PMID 23411577
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Coburn B, Morris AM, Tomlinson G, Detsky AS. Does this adult patient with suspected bacteremia require blood cultures? JAMA. 2012 Aug 1;308(5):502-11. doi: 10.1001/jama.2012.8262. PMID 22851117
- [Background] Gunsolus IL, Sweeney TE, Liesenfeld O, Ledeboer NA. Diagnosing and Managing Sepsis by Probing the Host Response to Infection: Advances, Opportunities, and Challenges. J Clin Microbiol. 2019 Jun 25;57(7):e00425-19. doi: 10.1128/JCM.00425-19. Print 2019 Jul. PMID 31043466
- [Background] Sweeney TE, Shidham A, Wong HR, Khatri P. A comprehensive time-course-based multicohort analysis of sepsis and sterile inflammation reveals a robust diagnostic gene set. Sci Transl Med. 2015 May 13;7(287):287ra71. doi: 10.1126/scitranslmed.aaa5993. PMID 25972003
- [Background] Sweeney TE, Wong HR, Khatri P. Robust classification of bacterial and viral infections via integrated host gene expression diagnostics. Sci Transl Med. 2016 Jul 6;8(346):346ra91. doi: 10.1126/scitranslmed.aaf7165. PMID 27384347
- [Background] Sweeney TE, Perumal TM, Henao R, Nichols M, Howrylak JA, Choi AM, Bermejo-Martin JF, Almansa R, Tamayo E, Davenport EE, Burnham KL, Hinds CJ, Knight JC, Woods CW, Kingsmore SF, Ginsburg GS, Wong HR, Parnell GP, Tang B, Moldawer LL, Moore FE, Omberg L, Khatri P, Tsalik EL, Mangravite LM, Langley RJ. A community approach to mortality prediction in sepsis via gene expression analysis. Nat Commun. 2018 Feb 15;9(1):694. doi: 10.1038/s41467-018-03078-2. PMID 29449546
- [Background] Sweeney TE, Khatri P. Benchmarking Sepsis Gene Expression Diagnostics Using Public Data. Crit Care Med. 2017 Jan;45(1):1-10. doi: 10.1097/CCM.0000000000002021. PMID 27681387
- [Derived] Whitfield NN, Hogan CA, Chenoweth J, Hansen J, Hsu EB, Humphries R, Mann E, May L, Michelson EA, Rothman R, Self WH, Smithline HA, Karita HCS, Steingrub JS, Swedien D, Weissman A, Wright DW, Liesenfeld O, Shapiro NI. A standardized protocol using clinical adjudication to define true infection status in patients presenting to the emergency department with suspected infections and/or sepsis. Diagn Microbiol Infect Dis. 2024 Sep;110(1):116382. doi: 10.1016/j.diagmicrobio.2024.116382. Epub 2024 May 31. PMID 38850687